CLINICAL TRIAL: NCT01112683
Title: A Sixteen-Week, Randomized, Double Blind, Placebo-Controlled Evaluation of the Efficacy, Tolerability and Safety of Memantine Hydrochloride on Enhancing the Cognitive Abilities of Young Adults With Down Syndrome
Brief Title: Efficacy and Safety of Memantine Hydrochloride in Enhancing the Cognitive Abilities of Young Adults With Down Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-0934; 06-0934 (Other: Colorado Multiple Institutional Review Board)
Record Dates: First submitted 2010-04-23; First posted 2010-04-28 (Estimated); Results first posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2012-12

CONDITIONS: Down Syndrome
Keywords: Down syndrome; Trisomy 21; Pattern Recognition Memory (PRM); Paired Associates Learning (PAL); California Verbal Learning Test (CVLT); Test of Reception of Grammar (TROG-II); Peabody Picture Vocabulary Test (PPVT-III); Scales of Independent Behavior revised (SIB-R)
MeSH Terms: conditions — Down Syndrome | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine (Experimental): The drug dosage will follow memantine's standard titration schedule (i.e., 5 mg/d week one, 5 mg/BID week two, 5 & 10 mg/d divided dose week three, 10mg/BID week four).
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): These are identically-looking pills to the ones in the Memantine Arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — The drug dosage will follow memantine's standard titration schedule (i.e., 5 mg/d week one, 5 mg/BID week two, 5 & 10 mg/d divided dose week three, 10mg/BID week four).
  Other Names: Memantine brand name in the USA is Namenda
  Arms: Memantine
Drug: Placebo — These are identically-looking pills to those in the Memantine Arm.
  Other Names: Sugar Pills
  Arms: Placebo

SUMMARY:
The purpose of this 16-week research study is to determine whether a drug called memantine hydrochloride (memantine) has the potential to help improve memory and other cognitive abilities of young adults with Down syndrome (DS). Memantine (Namenda®) is a drug approved by the Food and Drug Administration (FDA) for patients with moderate to severe Alzheimer-type dementia. About 40 persons of both genders with Down syndrome aged 18-32 years will take part in this study. This is a randomized and double blind study. This means that subjects will have a 50/50 chance of being assigned to receive either the memantine pills or placebo (inactive pills). Neither the study participants nor the research personnel will know who is receiving active medication or placebo. Based on memantine's mode of action, current knowledge on brain pathology in persons with Down syndrome, and some preclinical data on mouse models of Down syndrome, we hypothesize that memantine may improve test scores of young adults with Down Syndrome on memory tests targeted at the function of the brain structure called the hippocampus. This research project has three specific aims: 1) investigate whether memantine has the potential to improve test scores on hippocampus-dependent measures in young adults with Down syndrome; 2) investigate whether memantine has the potential to improve test scores by these subjects on other cognitive measures; 3) investigate whether memantine is well tolerated by these subjects.

DETAILED DESCRIPTION:
Down syndrome, which is the result of the trisomy of Chromosome 21, is the most common genetically defined cause of intellectual disabilities. The estimated number of people with Down syndrome in the United States is approximately 300,000, and this figure is expected to continue increasing due to projected increases in the life expectancy of people with Down syndrome. Although this population trend reflects improvements in the general health care of individuals with Down syndrome, there has not been a parallel progress in the understanding of the pathogenesis and potential treatment of the psychological and neurological components of this genetic condition. These include various degrees of intellectual disability, increased incidence of seizure disorder in relation to the general population, motor dysfunction (including hypotonia), abnormal oculomotor and vestibular functions, substantial visual deficits, a neuropathology indistinguishable from Alzheimer disease, and increased incidence of major depression and dementia in adults.

Over the last fifteen years, progress in the quantitative description of specific traits associated with Down syndrome, the availability of postnatal-viable aneuploid mouse models of Down syndrome, and our progressively more sophisticated knowledge of the human and mouse genomes have provided investigators in this field with a realistic opportunity to start bridging the gap between basic and clinical research.

Whereas individuals with Down syndrome maintain relatively high levels of social intelligence and procedural learning, they often suffer from grossly impaired declarative or explicit memory. Not surprisingly, brain structures associated with declarative memory, namely the hippocampal and parahippocampal regions of the medial temporal lobe, are the most severely affected in persons with Down syndrome. The nature of these deficits suggests that therapies targeting hippocampal function would be particularly efficacious in ameliorating the cognitive deficits seen in persons with Down syndrome and, consequently, would enhance their quality of life.

Glutamatergic neurons form the major excitatory system in the brain and play a pivotal role in many physiological functions. Apart from the physiological role of glutamate, excessive activation of its receptors can also evoke neuronal dysfunction and even damage/death. Cell death ascribed to an excessive activation of glutamate receptors has been termed 'excitotoxicity' and seems to occur in acute insults such as stroke and trauma, but it may be also associated with chronic neurodegenerative diseases such as Alzheimer disease. N-methyl-D-aspartate (NMDA) receptor (NMDAR) mediated glutamate excitotoxicity is thought to play a major role in Aβ-induced neuronal death. This idea is part of the foundation of the glutamatergic hypothesis (as opposed to the cholinergic hypothesis) for Alzheimer disease.

Memantine is an NMDAR antagonist that has been reported to be effective therapeutically in Alzheimer disease. It has been available in Germany as well as in most of the European Union for more than two decades. Recently, it has been approved for moderate to severe dementia in the US. The chemical name for memantine hydrochloride is 1-amino-3,5-dimethyladamantane hydrochloride. Memantine is an uncompetitive, moderate affinity, antagonist of NMDARs. It has been proposed that therapeutic doses of this drug inhibit the pathological effect of NMDAR activation while leaving unaffected NMDAR-mediated physiological processes involved in learning and memory. Recent preclinical data from the laboratory of this trial's P.I. on the mouse model for DS (Ts65Dn) have suggested a dysregulation of NMDAR activity in these animals and demonstrated improvement on learning and memory measures by the use of acute doses of memantine.

In all clinical trials so far, memantine was found safe and well tolerated. The tolerability of an NMDAR antagonist depends upon its affinity towards the receptors, unbinding kinetics, and voltage dependency. Memantine is thought to improve the fidelity of synaptic transmission. Such action is predicted to provide both neuroprotection and symptomatic restoration of synaptic plasticity by one and the same mechanism.

Recent open-label studies suggest that memantine may be clinically useful and well tolerated in young individuals with other conditions that produce cognitive disabilities, such as autism and attention deficit hyperactivity disorder (ADHD).

Because of the ubiquity of Alzheimer disease-type pathology in persons with Down syndrome, the preclinical findings consistent with dysregulation of NMDAR activity in mouse models of Down syndrome, the safety profile of memantine (which is superior to the AChE inhibitors that are already being tested in persons with Down syndrome), and the possibility that memantine may indeed delay the onset of Alzheimer disease-type pathology in young adults with Down syndrome, all the professionals involved with this project decided that a small-scale randomized controlled clinical trial was warranted at present.

We would like to emphasize that the goal of this study is to evaluate the efficacy, tolerability and safety of memantine hydrochloride in enhancing the cognitive abilities of young adults with Down syndrome aged 18-32 years. Therefore, the present investigation is a non-overlapping and complementary clinical trial to the randomized, placebo-controlled clinical trial on the efficacy and tolerability of memantine in preventing age-related cognitive deterioration and dementia in people with Down syndrome age 40 and over (http://www.clinicaltrials.gov/ct2/show/record/NCT00240760?term=down+syndrome&rank=15) currently being carried out by our colleagues in London.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with Down syndrome aged 18 to 32 years. The documented cytogenetic diagnosis should be either "Trisomy 21", or "Complete Unbalanced Translocation of the Chromosome 21".
* Female subjects must be documented not to be pregnant by serum testing at screening.
* Laboratory findings within normal limits or judged clinically insignificant at baseline.
* Vital signs must be within normal limits for their age. (Medically treated hypotension will be allowed.)
* Screening ECG must demonstrate predominately normal sinus rhythm. Minor abnormalities documented as clinically insignificant by the investigator will be allowed. (Subjects with clinically significant but stable ECG abnormalities may enter the trial only with the permission of the principal investigators.)
* Subjects and their authorized representative will provide written informed consent and assessment.
* Subjects who have been receiving any experimental drug for Down syndrome must undergo a washout (~ 30 days or five half-lives of the drug, whichever is longer).
* Sufficiently proficient in English to be capable of reliably completing study assessments.
* Able to swallow oral medication (crushing of tablets will not be permitted).
* Must have a reliable caregiver or family member who agrees to accompany the subject to all visits, provide information about the subject as required by this protocol, and ensure compliance with the medication schedule. The subject must have contact at least once a day with the caregiver.
* Generally good health and judged by the investigators to be able to fully participate in the trial.

Exclusion Criteria:

* Subjects weighing less than 40 kg.
* Any current psychiatric or neurologic diagnosis other than Down syndrome.
* Subjects who currently meet or have within the past five years met DSM-IV (Diagnostic and Statistical Manual) criteria for drug or alcohol abuse or dependence.
* Subjects who, in the judgment of the investigators, currently represent a significant suicide risk or who would require treatment with electro-convulsive therapy or with psychotropic drugs during the study or who have received treatment with a depot neuroleptic drug within 6 months of entering the study.
* Subjects who are hospitalized or residing in a skilled nursing facility or subjects who are anticipated to enter a nursing home within the next 6 months. (Subjects may reside in group homes of other residential settings where they do not require or receive skilled nursing.)
* Any active or clinically significant conditions affecting absorption, distribution or metabolism of the study drugs.
* Subjects with significant allergies to or other significant intolerance of memantine therapy, its ingredients, or with contraindications to memantine therapy as stated in the prescribing information.
* Subjects who are expected to require general anesthetics during the course of the study.
* History or presence of seizure disorder (less than 3 years) or encephalitis.
* History of malignant neoplasms treated within 3 years prior to study entry or where there is current evidence of recurrent or metastatic disease.
* Subjects with treated hypothyroidism must be on a stable dose of medication for at least 3 months prior to screening and have normal serum T-4 and thyroid-stimulating hormone at screening. Subjects with diabetes mellitus controlled by diet, oral medication or insulin must have an HbA1c of < 8.0% and random serum glucose value of < 170 mg/dl.
* Severe infections or a major surgical operation within 3 months prior to screening.
* History of persistent cognitive deficits immediately following head trauma.
* Subjects who have donated blood or blood products during the 30 days prior to screening who plan to donate blood while participating in the study or within four weeks after completion of the study.
* Subjects who may not be able to comply with the protocol or perform the outcomes measures due to significant hearing or visual impairment or other issues judged relevant by the investigators.

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Costa, MD, Ph.D, Principal Investigator — University of Colorado School of Medicine; Edward Goldson, MD, Study Director — Children's Hospital Colorado
Locations (1):
- The Children's Hospital, Aurora, Colorado, United States

REFERENCES:
- [Result] Boada R, Hutaff-Lee C, Schrader A, Weitzenkamp D, Benke TA, Goldson EJ, Costa AC. Antagonism of NMDA receptors as a potential treatment for Down syndrome: a pilot randomized controlled trial. Transl Psychiatry. 2012 Jul 17;2(7):e141. doi: 10.1038/tp.2012.66. PMID 22806212

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 42 persons with DS from both genders and between the ages of 18 and 32 were recruited from the community. Thirty nine participants had a cytogenetic diagnostic of trisomy 21 and 3 had complete unbalanced Robertsonian translocations involving a 14 and 21 homologue, leading to an additional chromosome 21.
Pre-assignment Details: Two screened subjects were excluded from the trial before assignment to groups: 1 due to an unrelated medical issue and 1 because we could not find age/gender matching subject. And 1 dropped from the trial after randomization due to personal reasons (death in the family).
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 19 | 20
Completed | 18 | 19
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 23.27 (3.52) | 22.60 (4.01) | 22.93 (3.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Changes in Neuropsychological Measures From Baseline to End of Study
Description: The hippocampus-dependent measures assessed in the present study are
  1. Pattern recognition memory* - Measures visual memory for non-namable designs; scale range in dataset 4-24; higher score indicates better performance
  2. Paired associates task* - Measures ability to learn visual associations between a picture and its location, and retention of this information over time; scale range in dataset 0-17; higher score indicates better performance
  3. California Verbal Learning Test (CVLT) - Children's Version** - Measures episodic verbal memory (sum of the items recalled over the 4 learning trials); scale range in dataset 0-35; higher score indicates better performance
  4. Rivermead Behavioral Memory Test-Children's version** - Measures episodic memory for visual information presented in context; scale range in dataset 1-20; higher score indicates better performance * used in power analysis calculation of sample size ** secondary measures associated with the primary hypothesis
Time Frame: These neuropsychological measures will be assessed one time 24 hours before the beginning of treatment and then a second time 16 weeks from the beginning of the treatment
Population: One participant dropped out of the study due to parent complaints of increased anxiety, and another was excluded from analyses due to side effects (increased and persistent anxiety) reported at study completion.
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 18 | 19
units on a scale
  Pattern recognition memory pre/post diff scores | -0.22 [-1.95 to 1.50] | -0.84 [-2.52 to 0.83]
  Paired associates task stages pre/post diff scores | 0.56 [-0.07 to 1.04] | 0 [-0.48 to 0.48]
  Paired associates task 1st trial pre/post diff | 0.39 [-1.05 to 1.83] | 0.68 [-0.72 to 2.09]
  CVLT Free Recall Total | 5.84 [3.47 to 8.21] | 2.53 [0.33 to 4.72]
  Rivermead Behavioral Memory Test | 1.3 [-0.56 to 3.16] | 0.79 [-0.98 to 2.56]
Statistical Analysis 1: Comparison: Memantine vs Placebo; 20 subjects per group were expected to provide 60% power to detect a between-group mean difference of 1.2 correct patterns (change from baseline to week 16) on the Paired Associates Learning and to provide 40% power to detect a between-group mean difference of 1.2 patterns recognized on the Pattern Recognition Memory. A two-sided test at type I error rate of 5% was used. Sample size incorporated an inflation factor of 20% to account for ineligibility of 10% of randomized participants; Test type: Superiority or Other; p = 0.403, Mixed Models Analysis; An alpha level of 0.05 or lower represents statistical significance, no correction was made for multiple comparisons to minimize type II errors

2. Secondary Outcome: Changes in Benchmark Neuropsychological Measures From Baseline to End of Study
Description: The neuropsychological benchmark measures assessed in this study are
  1. Peabody Picture Vocabulary Test-III (PPVT-III; range: -27.00 to 23.00)
  2. Test for the Reception of Grammar (TROG; range: -13.00 to 19.00)
  3. Verbal Fluency (from the Developmental Neuropsychological Assessment (NEPSY); range: -13.00 to 10.00)
  4. Recall of Digits (Differential Ability Scales; DAS; -50.00 to 59.00)
  5. Spatial working memory (SWM; part of the Cambridge Neuropsychological Test Automated Battery, or CANTAB; range: -9.00 to 8.00)
  6. Scales of Independent Behavior Revised (SIB-R; -12.00 to 26.00) All listed values represent differences in scores obtained at baseline subtracted from scores at 16-weeks of treatment. With the exception of the spatial working memory, for all measures, higher values represent better outcome. For the spatial working memory, lower values represent better outcome.
Time Frame: Benchmark neuropsychological measures will be assessed one time 24 hours before the beginning of treatment and then a second time 16 weeks from the beginning of the treatment
Population: These measures were not predicted to change due to memantine treatment. Measures of non-verbal reasoning, receptive language and vocabulary, short-term phonological memory, verbal and non-verbal working memory and adaptive/behavioral functioning were included.
Measure: Mean (90% Confidence Interval); unit: scores on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 18 | 19
scores on a scale
  Peabody Picture Vocabulary Test-III | 0.72 [-4.02 to 5.46] | -1.42 [-6.03 to 3.19]
  Test for the Reception of Grammar | 2.33 [-0.46 to 5.13] | -0.42 [-3.14 to 2.30]
  Verbal Fluency (from the NEPSY) | 0.78 [-1.18 to 2.74] | 0.21 [-1.69 to 2.12]
  Recall of Digits (DAS) | 5.39 [-3.88 to 14.66] | -7.47 [-16.50 to 1.55]
  Spatial working memory (strategy) | -0.06 [-1.70 to 1.59] | -1.47 [-3.07 to 0.12]
  Scales of Independent Behavior Revised (SIB-R) | 5.94 [2.02 to 9.85] | 4.88 [1.21 to 8.55]
Statistical Analysis 1: Comparison: Memantine vs Placebo; No power calculations were performed for the secondary measures; Test type: Superiority or Other; p = 0.371, Mixed Models Analysis — This P-Value refers to the SIB-R Broad independence score; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Changes of Safety and Tolerability Assessments at Baseline and End of Study
Description: Clinical history and physical examinations, electrocardiograms (ECGs), comprehensive clinical laboratory tests, and incidence of adverse event recording. The comprehensive clinical laboratory tests will include assessments of liver and kidney function, electrolytes, acid/base balance, and blood glucose and proteins. In addition, pregnancy tests will be performed on all female participants of childbearing potential.
Time Frame: Safety and tolerability assessments will be performed at three time points: 1) 1-7 days before beginning of treatment; 2) after 8 weeks from the beginning of the treatment; and 3) 16-17 weeks from the beginning of the treatment
Measure: Number; unit: participants
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 19 | 19
participants
  Increased anxiety | 2 | 0
  Transient dizziness | 1 | 0
  Echolalia | 1 | 0
  Androgenic alopecia | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the first day of treatment up to two weeks after the final week (16th week) of treatment, for a total of 18 weeks.
Arm/Group | Memantine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 3/19 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=19) | Placebo (N=19)
Androgenic alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Echolalia (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No